CLINICAL TRIAL: NCT00471159
Title: A Randomized Phase 2 Clinical Trial Of Docetaxel With Or Without PF-3512676 As First-Line Treatment Of Patients With Advanced Breast Cancer
Brief Title: A Study Of Docetaxel Or Docetaxel Plus PF-3512676 To Treat Patients With Advanced Breast Cancer.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501007
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; ProMune

INTERVENTIONS:
Drug: docetaxel
Drug: PF-3512676

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with docetaxel for the treatment of patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with confirmed advanced breast cancer.
* Patients with HER-2 negative disease with documented disease progression after (neo)adjuvant treatment with an anthracycline-based chemotherapy regimen.
* Patients with adequate general well-being, kidney and liver function.

Exclusion Criteria:

* Patients that have any condition that could affect patients safety, interfere with trial results, or makes the patient inappropriate for inclusion into study.
* Patients who have had prior chemotherapy for advanced breast cancer.
* Patients of child-bearing potential who are unwilling to use contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08

PRIMARY OUTCOMES:
Progression-free survival
Tumor assessment every 6 weeks until disease progression

SECONDARY OUTCOMES:
Overall objective response rate, duration of response, time to tumor progression - tumor assessment every 6 weeks until disease progression
Overall Survival - Patients will be followed for survival
Overall safety profile -Targeted questions to patients throughout study, Weekly blood sampling during treatment, every 3 weeks during follow-up, Urine sample every 3 weeks during treatment and follow-up
Changes in pain symptoms -Brief Pain Inventory questionnaire every 3 weeks during chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501007&StudyName=A%20Study%20Of%20Docetaxel%20Or%20Docetaxel%20Plus%20PF-3512676%20To%20Treat%20Patients%20With%20Advanced%20Breast%20Cancer.